CLINICAL TRIAL: NCT06434155
Title: Social History and Glaucoma Progression: The Effect of Body Mass Index, Tobacco, and Alcohol Consumption on the Rates of Structural Change in Patients With Open Angle Glaucoma
Brief Title: Social History and Glaucoma Progression
Acronym: OCT
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate Professor, Assiut University
Other Study IDs: 17200545
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Glaucoma Open-Angle
Keywords: Glaucoma; OCT
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Open Angle Glaucoma: 1. Patients older than 18 years of age with primary open-angle glaucoma (POAG)
  2. POAG diagnosed on the basis of IOP measurements more than 21 mmHg, Open angle on gonioscopy (Grade 3 or 4 on Schaffer grading system for angle width), glaucomatous visual field defects consistent with glaucomatous optic disc changes.
  3. Eyes with baseline macular and ONH OCT images and ONH photographs of adequate quality and r performed within 6 months of each other were selected

SUMMARY:
The objective of this study is to predict of glaucoma progression. By imaging of the retinal nerve fiber layer RNFL, optic nerve head (ONH) and macular measurements using spectral-domain OCT (SD-OCT) instruments

DETAILED DESCRIPTION:
Glaucoma is a multifactorial optic neuropathy characterized by structural damage of retinal ganglion cells (RGCs) and their axons that is associated with vision loss and may lead to irreversible blindness. Because glaucomatous damage is irreversible and effective treatment is available to halt further damage, glaucoma management should be optimized with precise micrometer-scale quantifications of ocular structures that improve detection of the disease and its progression. The introduction of OCT technology more than 20 years ago provided in vivo detailed visualization of the optic nerve head (ONH) and retina and enabled the quantitative evaluation of these tructures. Circumpapillary retinal nerve fiber layer (RNFL) thickness is a common OCT measurement that provides comprehensive evaluation of all RGCs in an eye as they converge into the ONH.

When measured with spectral-domain OCT, the RNFL has been shown to differentiate between healthy and glaucomatous eyes. The steady evolution of OCT technology has led to imaging with better resolution, higher scanning speeds, and advanced imaging patterns that has improved the reliability of OCT measurements and allowed for detection of minute changes that can improve the sensitivity of progression detection. Assessment of glaucoma progression usually is based on event or trend analysis. Event-based progression determines when a measurement exceeds a pre-established threshold for change from baseline. Trend-based analysis quantifies the rate of a parameter's progression over time.

ELIGIBILITY:
Inclusion Criteria:

* IOP measurements more than 21 mmHg
* Open angle on gonioscopy (Grade 3 or 4 on Schaffer grading system for angle width)
* Glaucomatous visual field defects consistent with glaucomatous optic disc changes.
* Eyes with baseline macular and ONH OCT images and ONH photograps

Exclusion Criteria:

* Participants with significant retinal disease.
* non-glaucomatous optic neuropathy.
* anomalous discs
* any retinal pathology.
* history of cataract or glaucoma surgery will not be exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age with primary open-angle glaucoma (OAG)
Sampling Method: Probability Sample
Enrollment: 1584 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
OCT structural parameters | 6 months
  RNFL in (um), ONH in (um), as well as the inner macula thickness (in um) using spectral domain OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt